CLINICAL TRIAL: NCT05374876
Title: Pilot Randomized Feasibility Trial Comparing Investigational Hand Therapy Intervention to Traditional Occupational Therapy Intervention to Prevent Chemotherapy-Induced Peripheral Neuropathy of the Hands in Patients Receiving Albumin Bound Paclitaxel + Gemcitabine Containing Combination Chemotherapy
Brief Title: Hand Therapy Intervention Versus Traditional Occupational Therapy to Prevent Chemotherapy Induced Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HonorHealth Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AX-CL-PANC-PI-003347
Record Dates: First submitted 2021-10-29; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Adenocarcinoma of Pancreas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational hand therapy (IHT)] intervention targeting the nervous system (Other)
  Interventions: Other: Hand Therapy Until CIPN
- Traditional occupational therapy intervention targeting compensatory strategies (TOT) (Other)
  Interventions: Other: Hand Therapy Until CIPN

INTERVENTIONS:
Other: Hand Therapy Until CIPN — Patient will participate until the time of onset of CIPN of the hands or through 84 days of treatment if no symptoms of CIPN.

SUMMARY:
A pilot randomized feasibility trial with a blinded evaluator.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) has a dose limiting effect which can greatly affect quality of life and often limits the amount of treatment patients can receive in treating their cancer. In the discipline of hand therapy, there is a science-based body of knowledge with effective protocols to treat neuropathies associated with injury and disease. These interventions have not been explored on patients with CIPN.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with adenocarcinoma of the pancreas who will receive chemotherapy with albumin bound paclitaxel plus gemcitabine containing combination
2. Patients who have no prior evidence of peripheral neuropathy of the hands
3. Age 18 years or older
4. Able to sit for minimum of 30 minutes for hand therapy sessions

Exclusion Criteria:

1. Patients who have received at least one dose of chemotherapy with albumin bound paclitaxel plus gemcitabine during the past 6 months
2. Patients taking duloxetine or gabapentin
3. History of peripheral neuropathy of the hands due to chemotherapy, diabetes, or other causes
4. Inability to sit for minimum of 30 minutes
5. Documented cognitive problems limiting ability to participate in hand therapy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Cutaneous Sensation | time of consent until the time of onset of CIPN of the hands or through 84 days of treatment
  measured by CTCAE Version 4

SECONDARY OUTCOMES:
Change in pain | time of consent until the time of onset of CIPN of the hands or through 84 days of treatment
  measured by visual analog scale
Change in moving touch sensation | time of consent until the time of onset of CIPN of the hands or through 84 days of treatment
  measured by TEN test
Change in innervation density | time of consent until the time of onset of CIPN of the hands or through 84 days of treatment
  measured by Two Point Discrimination Test
Change in pressure threshold sensation | time of consent until the time of onset of CIPN of the hands or through 84 days of treatment
  measured by monofilament test
Change in peripheral nerve tolerance at the thoracic level of the right and left arm | time of consent until the time of onset of CIPN of the hands or through 84 days of treatment
  measured by elevated arm stress test
Change in median nerve tolerance at the right and left volar wrist | time of consent until the time of onset of CIPN of the hands or through 84 days of treatment
  measured by Phalen's test
Change in ulnar nerve tolerance at the right and left elbow | time of consent until the time of onset of CIPN of the hands or through 84 days of treatment
  measured by elbow flexion test
Indication of irritability of the median and ulnar nerve at the right and left wrist | time of consent until the time of onset of CIPN of the hands or through 84 days of treatment
  measured by Tinel test

CONTACTS AND LOCATIONS:
Overall Officials: Gayle Jameson, Principal Investigator — HonorHealth Research Institute
Locations (1):
- HonorHealth Research Institute, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
Journal articles

REFERENCES:
- [Derived] Jameson GS, Cooper C, Snyder C, Buchanan SM, Strelish T, Shearon T, Von Hoff DD, Bay C, Hull L, Kaatz LA, Borazanci EH. Hand therapy interventions for the prevention of chemotherapy-induced peripheral neuropathy of the hands in patients with pancreatic cancer. Oncologist. 2024 Dec 6;29(12):1095-e1778. doi: 10.1093/oncolo/oyae285. PMID 39436905